CLINICAL TRIAL: NCT03178708
Title: The Implications of Amantadine Sulphate Usage in Spine Deformities Corrective Surgeries Patients as Regard Its Effect on the Duration of Wake up Test and Postoperative Opioid Consumption
Brief Title: Amantadine Sulphate Usage in Spine Deformities Corrective Surgeries Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IV amantadine
Record Dates: First submitted 2017-06-03; First posted 2017-06-07 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Spinal Curvatures
MeSH Terms: conditions — Spinal Curvatures | interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: the role of preoperative administration of Amantadine Sulphate on the duration of wake up test and postoperative opiod consumption in patients undergoing major spine deformities corrective surgeries.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A amantadine sulfate (Active Comparator): the patients will receive amantadine sulfate infusion using the dose 200 mg slowly I.V 3 hours prior to the surgery
  Interventions: Drug: Group A amantadine sulfate
- Group B ringer lactate (Placebo Comparator): the patients will receive 500 ml ringer lactate infusion slowly i.v 3 hours prior to surgery.
  Interventions: Other: Group B ringer lactate

INTERVENTIONS:
Drug: Group A amantadine sulfate — infusion solution for slowly intravenous application 3 hours preoperative
  Other Names: PK-Merz Infusion amantadine sulfate
  Arms: Group A amantadine sulfate
Other: Group B ringer lactate — infusion solution for intravenous application 3 hours preoperative
  Other Names: ringer lactate; Lactated ringer
  Arms: Group B ringer lactate

SUMMARY:
During the surgical procedure of scoliosis correction, large surgery extent and long-lasting strong nociceptive stimulation lead to postoperative pain formation of greater intensity compared with other orthopedic interventions. In these patients, duration of postoperative symptoms is longer, and may lead to persistent pain formation due to developing neuroplastic changes in the central nervous system.

DETAILED DESCRIPTION:
Instrumentation in correction operations for spinal deformities as vertebral fusion, congenital and traumatic scoliosis, carries a 0.5-5% risk of injuring the spinal cord during spinal surgery.

These complications are generally results of complex factors such as direct effects of compression on the spinal cord, distraction, the effects of spinal ischemia or arterial hypotension.

The purpose of the wake-up test is to monitor voluntary motor function of the lower limbs once the vertebrae have been instrumented and distracted. The depth of anesthesia is gradually lightened up to the point where patients are able to respond to verbal commands. As the voluntary movement of lower extremities is demonstrated, the depth of anesthesia is increased to complete the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Being candidate for spine deformity correction surgery(scoliosis and kyphosis )
2. Willing to participate in the study

Exclusion Criteria:

1. Patient refusal
2. Patients with chronic kidney, lungs,Gastrointestinal tract, liver, or cardiovascular diseases.
3. Pregnant or breastfeeding women.
4. Allergy to any of the study medications and taking medications that could significantly interact with amantadine (tramadol, atropine,antipsychotic medications)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
postoperative opioid consumption | 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

REFERENCES:
- [Result] Snijdelaar DG, Koren G, Katz J. Effects of perioperative oral amantadine on postoperative pain and morphine consumption in patients after radical prostatectomy: results of a preliminary study. Anesthesiology. 2004 Jan;100(1):134-41. doi: 10.1097/00000542-200401000-00022. PMID 14695734
- [Result] Eisenberg E, Pud D, Koltun L, Loven D. Effect of early administration of the N-methyl-d-aspartate receptor antagonist amantadine on the development of postmastectomy pain syndrome: a prospective pilot study. J Pain. 2007 Mar;8(3):223-9. doi: 10.1016/j.jpain.2006.08.003. Epub 2006 Sep 22. PMID 16996315
- [Result] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Result] Singla N, Rock A, Pavliv L. A multi-center, randomized, double-blind placebo-controlled trial of intravenous-ibuprofen (IV-ibuprofen) for treatment of pain in post-operative orthopedic adult patients. Pain Med. 2010 Aug;11(8):1284-93. doi: 10.1111/j.1526-4637.2010.00896.x. Epub 2010 Jun 30. PMID 20609131